CLINICAL TRIAL: NCT06711133
Title: Role of Multimodal Ultrasonography in Evaluation of Peripheral Neuropathy
Brief Title: Multimodal Ultrasound in Peripheral Neuropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Galal, Resident Doctor, Assiut University
Other Study IDs: Ultrasound in neuropathy
Record Dates: First submitted 2024-11-22; First posted 2024-12-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will enforce the role of ultrasound in early diagnosis and screening on peripheral neuropathy in comparison with other modalities.

DETAILED DESCRIPTION:
Each case will undergo informed Written consent and will be told the aim of the study including benefits, no harm from this procedure to the participants.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical symptoms of peripheral neuropathy

Exclusion Criteria:

* patients with unhealthy tissue texture to put on probe

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinical data of peripheral neuropathy who can cooperate to do the procedure not mentally retarded and healthy skin texture .
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
The Role of multimodal ultrasonography in evaluation of peripheral neuropathy | 3 years
  Enforce the role of ultrasound in screening and early detection of nerve affection in peripheral neuropathy in comparison with the traditional modalities as nerve biopsy and nerve conduction

REFERENCES:
- [Background] Telleman JA, Herraets IJ, Goedee HS, van Asseldonk JT, Visser LH. Ultrasound scanning in the diagnosis of peripheral neuropathies. Pract Neurol. 2021 Jun;21(3):186-195. doi: 10.1136/practneurol-2020-002645. Epub 2021 Feb 4. PMID 33541914